CLINICAL TRIAL: NCT06143371
Title: A Phase I (First-in-human) Randomized, Double-blind, Placebo Controlled Study to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of CAN10, an Anti-IL1RAP Monoclonal Antibody, in Healthy Subjects and in Subjects With Mild to Moderate Plaque Psoriasis.
Brief Title: A Study to Investigate the Safety and Tolerability of CAN10 Antibody in Healthy Subjects and in Subjects With Plaque Psoriasis.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAN10CLIN001; 2023-504450-35 (EudraCT Number)
Record Dates: First submitted 2023-11-16; First posted 2023-11-22 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Healthy; Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- CAN10 single ascending dose (Experimental): A single dose of CAN10 will be administered intravenously (IV) to healthy subjects.
  Interventions: Biological: CAN10
- CAN10 single ascending dose - placebo (Placebo Comparator): A single dose of matching placebo will be administered intravenously (IV) to healthy subjects.
  Interventions: Biological: CAN10 - Placebo
- CAN10 multiple ascending dose (Experimental): Multiple doses of CAN10 will be administered subcutaneously (SC) to subjects with mild to moderate plaque psoriasis
  Interventions: Biological: CAN10
- CAN10 multiple ascending dose - placebo (Placebo Comparator): Multiple doses of matching placebo will be administered subcutaneously (SC) to subjects with mild to moderate plaque psoriasis
  Interventions: Biological: CAN10 - Placebo

INTERVENTIONS:
Biological: CAN10 — Single dose intravenous or Multiple doses subcutaneously
  Arms: CAN10 multiple ascending dose; CAN10 single ascending dose
Biological: CAN10 - Placebo — Single dose intravenous or Multiple doses subcutaneously
  Arms: CAN10 multiple ascending dose - placebo; CAN10 single ascending dose - placebo

SUMMARY:
This is a first-in-human, randomized, double- blind, placebo-controlled, dose escalation study to investigate how different doses of CAN10 are tolerated, taken up by the body and how long CAN10 stays in the body. In the first part of the study, the single ascending dose (SAD) cohorts, CAN10 will be given as a single intravenous dose to healthy subjects. In the second part of the study, the multiple ascending dose (MAD) cohorts, CAN10 will be given as repeated subcutaneous doses to participants with mild to moderate plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 18 to 50 years of age (inclusive) at the time of signing informed consent.
* Body mass index (BMI) 18 to 30 kg/m2 (inclusive) and a weight between 50 to 100 kg (inclusive) at the time of screening
* Considered by the investigator to be in good general health as determined by medical history, clinical laboratory test results, vital sign measurements, 12-lead ECG results, and physical examination findings at screening.
* Female subjects of childbearing potential must use a highly effective method of birth control and have a negative pregnancy test at screening and before the first dose of study drug. Male subjects with female partners must agree to use a condom, and their female partners are recommended to use a highly effective method of birth control.

Additionally for subjects with plaque psoriasis only:

* A diagnosis of plaque psoriasis with Psoriasis Area Severity Index (PASI) score ≥3 to ≤15 and Physician Global Assessment (PGA) score ≥2 (mild) to <4 (moderate).
* No disease manifestation requiring systemic immunosuppressive therapy.

Exclusion Criteria:

* History or presence of:

  1. Severe allergy/hypersensitivity (subjects with mild pollen allergy can be included).
  2. Significant kidney, liver, or urologic disease.
  3. Clinically significant psychiatric disorders
  4. Tuberculosis (TB) infection or positive QuantiFERON TB Gold test
  5. Any other clinically significant disease or disorder which, in the opinion of the investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
* Clinically significant illness, medical/surgical procedure, or trauma within 4 weeks before the first dose of study drug.
* Ongoing opportunistic or systemic infections
* A positive test result for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus antigen or antibodies at screening.

Additionally for subjects with plaque psoriasis only:

* Psoriasis other than a plaque variant.
* Any sign of infection of any of the psoriatic lesions.
* Use of any of the following treatments within the indicated washout period before the first dose of study drug:

  1. 12 weeks or 5 half-lives (whichever is longer) for biologic agents known or expected to impact the course of psoriasis or its assessments.
  2. 12 weeks for oral retinoids
  3. 8 weeks for cyclosporin, interferon, methotrexate, other systemic immunosuppressive or immunomodulating agents, or psoralen plus ultraviolet A (UVA)
  4. 2 weeks for immunizations or drugs known to possibly worsen psoriasis, unless on a stable dose for >12 weeks
  5. 1 week for topical treatments: corticosteroids, immunomodulators, anthralin (dithranol), Vitamin D derivatives, retinoids, or coal tar (used on the body)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2023-08-21 (Actual); Primary Completion 2025-11-10 (Actual); Study Completion 2025-11-10 (Actual)

PRIMARY OUTCOMES:
To investigate the safety and tolerability of single and multiple ascending doses of CAN10 | From the day of the first dose until day 57 after the last dose
  Frequency, seriousness, and intensity of treatment-emergent adverse events (TEAEs) in subjects receiving single and multiple doses of CAN10

SECONDARY OUTCOMES:
Assessment of Area under plasma concentration time curve (AUC) from time 0 extrapolated to infinity (AUCinf) after single (IV) dosing | From the day of dosing (day 1) until day 57 after dosing
Assessment of AUC from time zero to last measurable serum concentration (AUClast) following single (IV) and multiple (SC) dosing | From the day of the first dose until day 57 after the last dose
Assessment of AUC from time 0 to 336 hours post dose (i.e., AUC over a 2-week interval) after multiple (SC) dosing on Day 36 (AUC0-336,MD) | From the last dose until 336 hours after the last dose
Assessment of the maximum observed concentration (Cmax) following single (IV) and multiple (SC) dosing | From the day of the first dose until day 57 after the last dose
Assessment of time to maximum observed serum concentration (Tmax) following single (IV) and multiple (SC) dosing | From the day of the first dose until day 57 after the last dose
Assessment of the terminal elimination rate constant (λz) following single (IV) and multiple (SC) dosing | From the day of the first dose until day 57 after the last dose
Assessment of the terminal halflife (t1/2) following single (IV) and multiple (SC) dosing | From the day of the first dose until day 57 after the last dose
Assessment of the total clearance (CL) following single (IV) dosing) | From the day of dosing (day 1) until day 57 after dosing
Assessment of the volume of distribution (Vd) following single (IV) dosing | From the day of dosing (day 1) until day 57 after dosing
Assessment of total clearance following extravascular administration (CL/F) following multiple (SC) dosing | From the day of the first dose until day 57 after the last dose
Assessment of volume of distribution following extravascular administration (Vd/F) following multiple (SC) dosing | From the day of the first dose until day 57 after the last dose

CONTACTS AND LOCATIONS:
Overall Officials: Manuela Casjens, MD, Principal Investigator — CRS Clinical Research Services Berlin GmbH
Locations (1):
- CRS Clinical Research Services Berlin GmbH, Berlin, Germany

REFERENCES:
- [Derived] Mulholland M, Depuydt MAC, Jakobsson G, Ljungcrantz I, Grentzmann A, To F, Bengtsson E, Jaensson Gyllenback E, Gronberg C, Rattik S, Liberg D, Schiopu A, Bjorkbacka H, Kuiper J, Bot I, Slutter B, Engelbertsen D. Interleukin-1 receptor accessory protein blockade limits the development of atherosclerosis and reduces plaque inflammation. Cardiovasc Res. 2024 May 7;120(6):581-595. doi: 10.1093/cvr/cvae046. PMID 38563353